CLINICAL TRIAL: NCT00288860
Title: Telephone Case Monitoring for Veterans With PTSD
Brief Title: Telephone Case Monitoring (TCM) for Veterans With Post-Traumatic Stress Disorder (PTSD)
Acronym: TCM-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEL 03-135
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: telemedicine; treatment compliance; mental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Patient Compliance; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone Monitoring (Experimental): Biweekly monitoring and support by telephone (up to 6 calls over 3 months) as augmentation to mental health care as usual.
  Interventions: Behavioral: Telephone monitoring; Other: Treatment-As-Usual
- Treatment-As-Usual (Active Comparator): Mental health Treatment As Usual, potentially including case management, pharmacotherapy, and individual and/or group psychotherapy.
  Interventions: Other: Treatment-As-Usual

INTERVENTIONS:
Behavioral: Telephone monitoring — Three months of biweekly telephone monitoring and support
  Arms: Telephone Monitoring
Other: Treatment-As-Usual — Outpatient mental health Treatment As Usual (psychotherapy and/or medications)

SUMMARY:
The purpose of this study is to test whether providing PTSD patients additional support by telephone (in addition to usual outpatient care) after they discharge from residential treatment improves those patients' outcomes and keeps them out of the hospital longer.

DETAILED DESCRIPTION:
Background: Poor compliance with aftercare may contribute to high rates of relapse and rehospitalization among Veterans who received residential treatment for posttraumatic stress disorder (PTSD). Telephone case monitoring has been shown to improve treatment adherence and reduced relapse among patients with chronic medical and substance use disorders, but has not been tested in PTSD patients.

Objectives: This multisite randomized controlled trial tested whether augmenting usual aftercare with telephone monitoring improved resulted in 1) improved clinical outcomes (less violence, substance use, and PTSD symptoms; 2) longer time to rehospitalization; 3) better compliance with aftercare in the year after discharge from residential treatment for PTSD.

Methods: This trial recruited 837 subjects from 6 PTSD residential treatment programs at 5 VA medical centers, 94.7% of the 884 projected. Patients who completed at least 14 days of residential PTSD treatment and discharged to VA outpatient care were eligible to participate. Subjects were randomized to usual aftercare care (n = 425) or usual aftercare plus biweekly telephone case monitoring calls during the first three months after discharge (n = 412). Telephone case monitors assessed current problems, encouraged treatment adherence, provided problem-solving support, and alerted providers to emergent care needs. Patient self-report measures of psychiatric symptoms, substance use, and violence were obtained at intake to residential treatment and 4 months (69% completion rate) and 12 months (64% completion rate) after discharge. Retention was lower than the investigators' planned 70% to 75% rate due to difficulty locating some patients who moved (even their collateral informants did not know where they were) and 45 participants asking to discontinue due to lack of time (n = 10), general dissatisfaction with VA (n = 6), distress during phone calls (n = 5), dissatisfaction with compensation (n = 1), or no specified reason (n = 24). Treatment utilization data was obtained from the VA National Patient Care Database.

Intent-to-treat analyses used mixed modeling to compare clinical outcomes in the telephone monitoring and usual care groups and 4 and 12 months after discharge. Survival analysis was used to compare conditions on time to rehospitalization. Having a slightly smaller-than-intended sample size resulted in modest reductions in statistical power, e.g., power to detect the expected d = .25 effect on PTSD outcomes was reduced from about 90% to 82%, and power to detect the anticipated W = .105 difference in rehospitalization rates was reduced from 88% to 85%. Secondary analyses assessed whether differences in outcomes between the telephone case monitoring and usual care groups were mediated by attending more outpatient visits and completing more medication refills. Exploratory analyses examined whether the effect of telephone support on the clinical outcome measures, number of treatment visits, and medication refills was moderated by number of outpatient mental health visits in the prior year, distance from clinic, treatment expectancies, therapeutic alliance, or co-occurring substance use problems.

Status: Enrollment, intervention, data collection, and primary analyses are completed. Primary results have been published in Psychiatric Services (Rosen, Tiet, Harris et al., 2013) and two secondary papers have been published in the Journal of Traumatic Stress (Belsher, Tiet, Garvert, & Rosen, 2012; Rosen, Adler, & Tiet, 2013).

A CDMRP-funded study extending this approach to PTSD outpatients at the Durham, Puget Sound and Palo Alto VA medical centers has recently been completed. Initial results of that second trial suggest that telephone care management improved treatment attendance but had weak effects on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PTSD diagnosis entering PTSD residential treatment with an intended length of stay of 15 days or longer (patients in brief evaluation or acute stabilization tracks will not be included, as their discharge plan may include readmission to residential treatment within a few months).

Exclusion Criteria:

1. Patients discharging from residential treatment within four days of admission(insufficient time to consent and assess them);
2. Active Duty military personnel;
3. Patients transferred from residential care to an inpatient medical unit due to emergent medical problems;
4. Patients with traumatic brain injury or other organic impairment that compromises capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2006-10; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig S. Rosen, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (5):
- United States (5):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - VA Medical Center, Battle Creek, Battle Creek, Michigan
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - VA Medical Center, Coatesville, Coatesville, Pennsylvania
  - VA Puget Sound Health Care System, Tacoma, Tacoma, Washington

REFERENCES:
- [Result] Rosen CS, Tiet QQ, Harris AH, Julian TF, McKay JR, Moore WM, Owen RR, Rogers S, Rosito O, Smith DE, Smith MW, Schnurr PP. Telephone monitoring and support after discharge from residential PTSD treatment: a randomized controlled trial. Psychiatr Serv. 2013 Jan;64(1):13-20. doi: 10.1176/appi.ps.201200142. PMID 23117443
- [Result] Belsher BE, Tiet QQ, Garvert DW, Rosen CS. Compensation and treatment: disability benefits and outcomes of U.S. veterans receiving residential PTSD treatment. J Trauma Stress. 2012 Oct;25(5):494-502. doi: 10.1002/jts.21747. Epub 2012 Oct 9. PMID 23047625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans entering treatment in five 30-to-90 day residential treatment programs for posttraumatic stress disorder
Pre-assignment Details: 926 patients were initially consented into the study. 6 withdrew prior to randomization, and 83 met exclusion criteria after being consent (usually because they were discharged to another inpatient program, not to outpatient care). This left 837 subjects to be randomized.
Groups:
- Telephone Monitoring: Telephone monitoring as augmentation to treatment as usual
  Telephone case monitoring: Three months of biweekly telephone monitoring and support in addition to usual outpatient mental health care (psychotherapy and/or medications)
- Treatment-As-Usual: Treatment as usual
  Treatment as Usual Control: Usual outpatient mental health care (psychotherapy and/or medications)
Period: Overall Study
Arm/Group | Telephone Monitoring | Treatment-As-Usual
Started | 412 | 425
Completed Intake Survey | 408 | 417
Completed 4 Month fu Survey | 275 | 299
Completed 12 Month fu Survey | 257 | 281
Completed | 310 (310 completed either 4 or 12 month survey. Used all with intake (n = 408) in intent-to-treat.) | 328 (328 completed 4 or 12 month survey. Used all with intake (n=417) in intent to treat.)
Not Completed | 102 | 97
Not completed — Did not complete intake | 4 | 8
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 20 | 15
Not completed — Lost to Follow-up | 74 | 71

BASELINE CHARACTERISTICS:
Population: Veterans entering residential treatment for posttraumatic stress disorder.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Monitoring | Treatment-As-Usual | Total
Number analyzed (Participants) | 412 | 425 | 837
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (0.62) | 49.9 (0.86) | 50.0 (0.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 57 | 112
  Male | 357 | 368 | 725
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 263 | 256 | 519
  African American | 87 | 93 | 180
  Asian American | 2 | 0 | 2
  Native American | 11 | 8 | 19
  Pacific Islander | 2 | 2 | 4
  Latino | 19 | 26 | 45
  Other | 22 | 28 | 50
  Race/ethnicity missing | 6 | 12 | 18
Iraq or Afghanistan veteran [Number; unit: participants]
  Iraq/Afghanistan veteran | 114 | 114 | 228
  Served prior to current Iraq/Afghanistan conflicts | 298 | 311 | 609

OUTCOME MEASURES:

1. Primary Outcome: Aggressive Behavior; Alcohol Misuse; Drug Misuse; PTSD Symptoms
Description: Higher scores are worse outcomes on all four measures:
  Aggressive behavior (scale from 0-6 types of violent behavior than past four months) - adapted from conflict tactics scale Alcohol problems: Addiction Severity Index Alcohol composite (ranges from 0 to 1) Drug problems: Addiction Severity Index Drug composite (ranges from 0 to 1) PTSD symptoms: DSM IV PTSD Checklist (ranges from 17 to 85)
Time Frame: 12 months post-discharge (8 months post intervention)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Treatment as Usual: Treatment as usual
  Treatment as Usual Control: Usual outpatient mental health care (psychotherapy and/or medications)
Arm/Group | Telephone Monitoring | Treatment as Usual
Number analyzed (Participants) | 412 | 425
Scores on a scale
  PTSD Symptoms (PTSD Checklist) | 63.9 (13.0) | 63.4 (12.5)
  Aggressive Behavior | 3.0 (2.2) | 3.1 (2.2)
  Alcohol Problems (ASI) | 0.15 (0.19) | 0.17 (0.19)
  Drug Problems (ASI) | 0.05 (0.09) | 0.05 (0.08)

2. Secondary Outcome: Depressive Symptoms, Subjective Quality of Life
Description: Depression: Center for Epidemiological Studies Scale (ranges from 0 to 60, with higher scores indicating worse depression) Quality of Life: Scale from the Veterans Affairs Military Stress Treatment Assessment (scores range from 1 to 7, with higher scores indicating better quality of life)
Time Frame: 12 months post-discharge (8 months post intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Monitoring | Treatment-As-Usual
Number analyzed (Participants) | 408 | 417
units on a scale
  Depression (CES-D) | 38.0 (10.1) | 38.4 (10.4)
  Quality of Life | 3.3 (1.1) | 3.3 (1.1)

3. Primary Outcome: Rehospitalization
Description: Number of patients with psychiatric hospitalization within 12 months of discharge from PTSD program
Time Frame: 12 months post discharge
Measure: Number; unit: participants
Groups:
- Telephone Monitoring: Biweekly monitoring and support by telephone (up to 6 calls over 3 months) as augmentation to mental health care as usual.
  Telephone monitoring: Three months of biweekly telephone monitoring and support
  TAU: Outpatient mental health Treatment As Usual (psychotherapy and/or medications)
- Treatment-As-Usual: Mental health Treatment As Usual, potentially including case management, pharmacotherapy, and individual and/or group psychotherapy.
  TAU: Outpatient mental health Treatment As Usual (psychotherapy and/or medications)
Arm/Group | Telephone Monitoring | Treatment-As-Usual
Number analyzed (Participants) | 412 | 425
participants | 45 | 55

ADVERSE EVENTS:
Time Frame: 12 months
Description: Serious adverse events (primarily death and hospitalizations) were tracked for both arms of the study.
Arm/Group | Telephone Monitoring | Treatment-As-Usual
Serious Adverse Events (participants affected / at risk) | 16/412 | 12/425
Other Adverse Events (participants affected / at risk) | 1/412 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Monitoring (N=412) | Treatment-As-Usual (N=425)
Death doe to causes not known (Social circumstances) | 4 (4) | 3 (3) — Cause of death not specified
Hospitalization for overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hospitalization for cardiology or chest pain (Cardiac disorders) | 2 (2) | 1 (1)
Scheduled laminotomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Psychiatric Hospitalization (Psychiatric disorders) | 10 (10) | 7 (7)
hospitalized for cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
kidney failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Arrest or incarceration (Social circumstances) | 2 (2) | 1 (1)
Admitted to nursing home - reason not known (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Monitoring (N=412) | Treatment-As-Usual (N=0)
Phone telephone care management upsetting (Psychiatric disorders) | 1 (1) | 0 (0) — Telephone Monitoring arm: Participant was sufficiently upset by telephone calls to ask to discontinue intervention. Treatment as Usual arm: Not applicable (0 subjects at risk) because did not receive this intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No